CLINICAL TRIAL: NCT07330804
Title: STUDY OF THE DOUBLE POLYMORPHISM (THR 555ILE) AND (GLU568PRO) OF THE CORIN GENE AS A RISK FACTOR FOR ARTERIAL HYPERTENSION IN A POPULATION OF AFRICAN DESCENT IN GUADELOUPE
Acronym: HTAG-CORIN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de la Guadeloupe (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: PAP_RIPH2_2024/01
Record Dates: First submitted 2025-04-28; First posted 2026-01-09 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-01

CONDITIONS: High Blood Pressure
Keywords: double polymorphisme; Corin; natriuretic peptide; biomarker; Afro Caribbean
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- cases (Other): Patients, considering themselves to be of Afro-Caribbean origin with hypertension, treated for hypertension or diagnosed as carrying hypertension according to HAS recommendations (Prise en charge de l'Hypertension artérielle de l'adulte, sept 2016): "elevation of blood pressure (BP), including systolic blood pressure (SBP) ≥140 mmHg and/or diastolic blood pressure (DBP) ≥ 90 mmHg" measured in the doctor's office and confirmed over several consultations on the day of inclusion.
  The diagnosis of hypertension can also be made by self-measurement over 3 days (mean PAS >135 mmHg and/or PAS> 85 mmHg) or by ABPM (Ambulatory Blood Pressure Monitoring: Holter Tensionnel) with PAS >135 mmHg and/or PAD >85 mmHg for the daytime period (awake); PAS>120 mmHg and/or PAD> 70 mmHg for the nighttime period (asleep).
  In the case of hypertension, mean PAS > 130 mmHg and PAD > 80 mmHg. ESC/ESH 2018 recommendations
  Interventions: Diagnostic Test: double polymorphism
- Controls (Other): Patients who consider themselves to be of Afro-Caribbean origin, of the same sex and ± 5 years of age as the cases, with no diagnosis of hypertension. Controls will be recruited by the same physicians who included a person with hypertension, but consulting for any other symptoms.
  Interventions: Diagnostic Test: double polymorphism

INTERVENTIONS:
Diagnostic Test: double polymorphism — diagnostic test
  Other Names: cases

SUMMARY:
Cardiovascular disease (CVD) mortality is the leading cause of death in high-income countries (particularly the United States), accounting for 23.1% of all deaths It has been established over several decades that hypertension disproportionately affects African Americans, compared with Americans of European descent:Hypertension occurs more often, at an earlier age , with greater severity , and is associated with an approximately 3-fold higher probability of death .There is also poorer control of hypertension despit e similar treatment In African Americans, CVD morbidity and mortality are compounded by the higher prevalence of T2DM, obesity, CKD, stroke, and heart failure . Despite advances in the identification of risk factors and the availability of effective treatment in hypertension, CVD disparities, persist among African Americans and are expected to increase in the future, particularly in younger age groups. Although various environmental and social factors certainly contribute to these disparities, a genetic basis, involving numerous "candidate" genes, is most often asserted in the literature . One of these is the Corin gene (Pan et al, 2002) which codes for the Corin protein.The latter plays a pivotal role in cardiometabolic pathophysiology through its role in the activation of natriuretic peptides .Natriuretic peptides (ANP and BNP) have a major role in the regulation of blood pressure through their vasodilatory and diuretic action. They have a lusotropic action, inhibit the renin angiotensin system, and are involved in energy metabolism (increased lipolysis and insulin secretion). They also have an anti-fibrotic, anti-proliferative, anti-inflammatory and anti-thrombotic action.The Corin gene of 244109pb has many variants that produce an inefficient protein with the corollary of the appearance of metabolic and cardiovascular pathologies in the first rank of which the HTA, the cardiac insufficiency and the renal insufficiency .Recently, a double polymorphism of the Corin gene consisting of 2 SNPs (single nucleotide polymorphisms) on the same allele of the Corin gene (I555/P568) has been reported. This allele is present in the heterozygous state in 12% of African Americans but is extremely rare in Americans of European descent (<0.5%).This double polymorphism (I555/P568) has been shown to be responsible for an approximately 70% reduction in the ability of the mutated Corin protein to convert proANP or proBNP to the active form. In addition, the I555(P568) allele of Corin protein is associated with an increased risk of hypertension and concentric cardiac hypertrophy The corin allele (I555/P568) is reported to be associated with poorer response to validated heart failure therapy and a higher risk of death or hospitalization for heart failure .

In Guadeloupe, where the population is predominantly of African descent.Cardiovascular disease is the leading cause of mortality.The prevalence of hypertension is 39% and more than 50% after 50 years of age . It has increased by 10% in 10 years in Guadeloupe. In France, where the prevalence of hypertension is 31%, it has increased by only 5% over the same period.

Heart failure is the main cause of admission to the cardiological emergency room of the University Hospital (49%) with a mortality of 37% at 6 months. Hypertension is the first risk factor associated with heart failure (80%).To date, there are no studies on corin gene polymorphisms in Guadeloupe. Following the example of work already done in the African American population, we propose to study the role of the double polymorphism (I555/P568) in the determinism of hypertension in the population of African descent in Guadeloupe.

ELIGIBILITY:
Inclusion Criteria:

Case inclusion criteria

* Persons affiliated with or benefiting from a social security plan;
* Over 18 years of age;
* Considering themselves to be of Afro-Caribbean descent;
* Having given their free, informed, written and signed consent (at the latest on the day of inclusion and before any examination required by the research);
* Treated for hypertension or presenting with hypertension according to recommendations: elevated blood pressure (BP), including systolic blood pressure (SBP) ≥140 mmHg and/or diastolic blood pressure (DBP) ≥ 90 mmHg measured in the physician's office and confirmed over several visits on the day of inclusion or diagnosis made by ABPM or self-measurement.

Control inclusion criteria:

* Individuals affiliated with or benefiting from a social security plan;
* Over 18 years of age;
* Patients who consider themselves of Afro-Caribbean origin, of the same sex as the cases and ± 5 years of age, not treated for hypertension and not presenting with hypertension according to the HAS recommendations on the day of the inclusion visit. Controls will be recruited by the same GPs who included a person with hypertension, consulting for any other symptom
* Having given their free, informed, written and signed consent (at the latest on the day of inclusion and before any examination required by the research);

Exclusion Criteria:

* Minors; Pregnant or breastfeeding women; Protected persons, or persons under court protection; Refusal to participate. Patients unable to come to the laboratory

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 370 (Estimated)
Dates: Start 2025-01-16 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
double polymorphism | At day 15
  1. Genotyping by capillary electrophoresis (Sanger sequencing):
  2. Genotyping using the allelic discrimination method

SECONDARY OUTCOMES:
heart failure | At inclusion
  Frequency of heart failure in cases and controls
Renal failure | At Day 15
  Frequency of renal failure in cases and
natriuretic peptid (NT PRO BNP) | At Day 15
  natriuretic peptid assay in cases and controls
créatinine clearance | At Day 15
  creatinine clearance in MDRD in cases and controls
Fasting blood glucose | At Day 15
  Hb1AC measurement
Cholesterolemia | At Day 15
  measurement
triglyceridemia | At Day 15
  measurement
Body Mass Index | At inclusion
  Body mass Index calculation measurement in cases and controls
waist | At inclusion
  waist circumference measurement in cases and controls
Left ventricular ejection fraction (LVEF)_systolic function in Simpson | At 3 months for case, 12 months control
  pourcentage
ECG measurements Cornell | At inclusion, or month 3 for case and month 12 for control
  mV
diastolic function E/ea ratio | At inclusion, or month 3 for case and month 12 for control
  ratio
parietal thickness | At inclusion, or month 3 for case and month 12 for control
  mm
left atrial size and volume | At inclusion, or month 3 for case and month 12 for control
  ml
ECG measurement Lewis | At inclusion, or month 3 for case and month 12 for control
  mV
ECG measurement Sokolow-Lyon | At inclusion, or month 3 for case and month 12 for control
  mV
ECG measurment Siegel | At inclusion, or month 3 for case and month 12 for control
  mV
ECG measurment Roberts | At inclusion, or month 3 for case and month 12 for control
  mV

CONTACTS AND LOCATIONS:
Locations (2):
- Guadeloupe (2):
  - Medical practice KERIB, Petit-Bourg
  - Toncoeurtonka, Petit-Canal